CLINICAL TRIAL: NCT03001999
Title: A Novel Psychological-behavioral Intervention to Improve Activity in Type 2 Diabetes: Proof-of-concept Trial
Brief Title: Boosting Emotions & Happiness in Outpatients Living With Diabetes: Phase I
Acronym: BEHOLD-16
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Jeff C. Huffman, MD, Associate Professor in Psychiatry, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016P002523
Record Dates: First submitted 2016-12-16; First posted 2016-12-23 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Type 2 Diabetes; Emotions; Patient Compliance
Keywords: Diabetes; Positive Psychology; Physical Activity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Patient Compliance; Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention Arm (Experimental): Participants will all undergo a 16-week PP-MI health behavior intervention.
  Interventions: Behavioral: PP-MI health behavior intervention

INTERVENTIONS:
Behavioral: PP-MI health behavior intervention — The positive psychology exercises include 3 modules:
  Gratitude-based activities, Strength-based activities, and Meaning-based activities. Various goal setting exercises will appear in each of the 14 study sessions.

SUMMARY:
The focus of this study is to examine the feasibility, acceptability, and preliminary impact of a customized, combined positive psychology and motivational interviewing (PP-MI) health behavior intervention in a group of patients with type 2 diabetes (T2D).

DETAILED DESCRIPTION:
The investigators are proposing a study that will specifically and innovatively focus on the development of a novel positive psychology intervention that is adapted for patients with T2D. The MGH Diabetes Center and MGH primary care clinics will serve as the source of subjects for the study, with patients who have a diagnosis of T2D serving as potential subjects. The investigators will enroll 12 T2D patients, who will take part in an 16-week PP-MI health behavior intervention.

In this project, the investigators plan to do the following:

1. Test a 16-week, telephone-delivered health behavior intervention utilizing PP exercises and systematic goal-setting in a brief, non-randomized, proof-of concept trial (N=12).
2. Determine whether this initial intervention is feasible in a small cohort of T2D patients.
3. Explore potential benefits of the intervention on outcomes of interest (e.g., optimism, positive affect).

Baseline information about enrolled participants will be obtained from the patients, care providers, and the electronic medical record as required for characterization of the population. This information will include data regarding medical history (type 2 diabetes mellitus), current medical variables (conditions affecting physical activity), medications, and sociodemographic data (age, gender, race/ethnicity, living alone).

Participants will undergo an initial screening visit during which they will meet with study staff in person. At this visit, study eligibility will be confirmed, and eligible and willing participants will be enrolled. Following enrollment, participants will complete self-report measures, and nurses in the Translational and Clinical Research Center will collect vital signs and draw blood for A1c. To ensure that participants have low baseline physical activity, they will then take home and wear accelerometers for 1 week.

Participants will undergo a second in-person visit to confirm that participants are eligible to complete the program and--if so--to initiate the program. During this session, A1c and accelerometer data will be reviewed. Participants will be required to have an A1c value between 6.5% and 9%, unless they have had an eligible A1c level in the past 6 months, in which case their current A1c may be between 6% and 9.5%. Furthermore, participants must have low physical activity (< 75 minutes of moderate or vigorous physical activity over the past week, measured by accelerometer) to continue in the program. Upon confirmation of eligibility, participants will begin the study intervention.

During this second in-person visit, participants will receive a PP-MI treatment manual. For each session, a PP exercise will be described in the manual, with instructions and space to write about the exercise and its effects. Next, an MI section will outline specific MI-based topics (e.g., pros/cons, managing slips) and facilitate physical activity goal-setting. Interventionists will complete PP exercise 1 and MI session 1 together with participants to aid engagement. Interventionists will also explain/assign PP exercise 2 and discuss an MI-based activity goal matched to participants' stage of change and medical recommendations (and assign activity tracking).

Participants will complete the remaining sessions (14 in total) by phone over the next 16 weeks. Phone sessions will last for approximately 30 minutes, with PP and physical activity assignments completed between phone sessions. PP and MI components will be delivered stepwise within sessions (rather than intertwined) based on our experience, participant feedback, and pilot work. If a week is missed, the session will not be skipped, but rather the intervention will be completed sequentially (with participants who miss weeks then missing the final sessions), with the exception of the final visit, which skip to Planning for the Future in all cases.

Participants will undergo an in-person follow-up assessment at 16 weeks. At this session, participants will repeat self-report assessments that were administered at baseline. Vital signs and a blood sample will again be collected at this final in-person visit. Finally, prior to this assessment, participants will wear an accelerometer for an additional 7 days to measure moderate or vigorous physical activity. The investigators will allow a window of 3 weeks, to allow flexibility of scheduling such in-person appointments in Boston (and to allow coordination with other medical visits at MGH) while maintaining integrity of study findings.

ELIGIBILITY:
Inclusion Criteria:

* T2D. Eligible patients will be diagnosed with T2D, with diagnosis for at least 1 year, confirmed by their diabetes clinician or medical record review. Consistent with American Diabetes Association (ADA) criteria for T2D, participants must have HbA1c [A1C] of at least 6.5% within the last 6 months. The investigators will exclude patients with A1C>9% given that patients in this range will likely have more extreme nonadherence and/or require ongoing treatment adjustment, increasing the heterogeneity of this sample for this pilot project. If patients appear otherwise eligible, but do not have an A1C value within 6 months, they will be required to have a baseline A1C value of 6.5-9%.
* Low physical activity. The investigators will define low physical activity as ≤75 minutes/week of MVPA (representing ≤40% of ADA recommendations for moderate or greater intensity aerobic physical activity totaling 150 minutes per week). This cutoff allows adequate room for improvement on this key outcome. As an initial screen, the investigators will use a modified version of the International Physical Activity Questionnaire (IPAQ) which has been extensively used/validated in medical cohorts, including T2D. Patients will complete the modified IPAQ regarding their activity in the past week (or a typical week, if the past 7 days atypical) to assess number of minutes spent performing MVPA. Patients reporting ≤60 minutes/week of MVPA will then wear accelerometers for 7 days to confirm low physical activity.
* Prescribed an oral glucose-lowering drug or choosing lifestyle interventions (diet and exercise) to manage T2D. To be eligible, patients must be prescribed a stable glucose-lowering medication regimen (or stable plan for control with diet/exercise alone) for at least 3 months with no anticipated adjustment. Including those whose T2D is managed by diet and exercise alone will allow inclusion of participants who may have high likelihood of engagement in a behavioral intervention. The investigators will exclude patients taking insulin to reduce heterogeneity of T2D severity in this initial trial.

Exclusion Criteria:

* Cognitive impairment precluding consent or meaningful participation, assessed using a six-item screen developed for this purpose.
* Lack of phone availability.
* Inability to read/write in English.
* Additional medical conditions (e.g., severe arthritis, chronic pulmonary obstructive disease, class III or IV heart failure) that preclude physical activity.
* Enrollment in mind-body programs, lifestyle intervention programs (e.g., cardiac rehabilitation), or other clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment procedures | Change between baseline and 16 weeks
  Feasibility will be measured by rates of enrollment per month.
Feasibility of study procedures | Change between baseline and 16 weeks
  Feasibility will also be measured by rates of dropout (%of total enrolled).

SECONDARY OUTCOMES:
Feasibility of intervention exercises | Change between baseline and 16 weeks
  Feasibility of intervention exercises will be measured by rates of completion of exercises.
Ease of intervention | Change between baseline and 16 weeks
  Ease of the intervention will also be measured by patient rating of the ease of PP-MI sessions on a 10-point Likert scale.
Utility of intervention | Change between baseline and 16 weeks
  Utility of the intervention will also be measured by patient rating of the utility of PP-MI sessions on a 10-point Likert scale.
Moderate-Vigorous Physical activity | Change between baseline and 16 weeks
  Physical activity changes will be measured by MVPA in mean minutes per day.
Sedentary Time | Change between baseline and 16 weeks
  Sedentary time will be measured in mean minutes per day.
Changes in PANAS Scores | Baseline and 16 weeks
  The positive affect items on the Positive and Negative Affect Schedule (PANAS), a well-validated scale used in other intervention trials and in patients with HF, will be used to measure positive affect.
Changes in LOT-R Scores | Baseline and 16 weeks
  Life Orientation Test-Revised is a well-validated 6-item instrument used to measure dispositional optimism.
Changes in HADS Scores | Baseline and 16 weeks
  The Hospital Anxiety and Depression Scale will be used to measure depression and anxiety. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients.
Changes in SEE Scores | Baseline and 16 weeks
  The Self-Efficacy for Exercise scale will be used to identify factors that may affect participation in exercise.
Changes in RS Scores | Baseline and 16 weeks
  The Resilience Scale will be used to examine the impact of the intervention on resilience.
Changes in MSPSS Scores | Baseline and 16 weeks
  The Multidimensional Scale of Perceived Social Support will be used to assess the intervention's impact on perceived social support.
Changes in SDSCA Scores | Baseline and 16 weeks
  The Summary of Diabetes Self-Care Activities will be used to evaluate overall diabetes self-care (e.g., diet, medication, foot care).

OTHER OUTCOMES:
Changes in T2D medication adherence | Baseline and 16 weeks
  The investigators will use a %-based self-report measure to gain estimates of T2D medication adherence.
Changes in IPAQ Scores | Baseline and 16 weeks
  The International Physical Activity Questionnaires will be used to assess changes in physical activity over the course of the study.
Changes in PF-20 Scores | Baseline and 16 weeks
  The 20-item short form of the Patient-Reported Outcomes Measurement Information System (PROMIS) will be used to assess physical function.
Changes in PDI Scores | Baseline and 16 weeks
  The Pain Disability Index will be used to assess pain-related disability.
Changes in Audit-C Questionnaire Responses | Baseline and 16 weeks
  This questionnaire will be used to assess changes in alcohol consumption over the course of the study.
Changes in Cigarette Use Questionnaire | Baseline and 16 weeks
  This questionnaire will be used to assess changes in cigarette use over the course of the study.
Blood pressure | Baseline and 16 weeks
Weight | Baseline and 16 weeks
Body mass index (BMI) | Baseline and 16 weeks
Hemoglobin A1c | Baseline and 16 weeks
  Patients will have their blood drawn at baseline and 16 weeks so that the investigators can obtain and assess their A1C level over the course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff C Huffman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Millstein RA, Golden J, Healy BC, Amonoo HL, Harnedy LE, Carrillo A, Celano CM, Huffman JC. Latent growth curve modeling of physical activity trajectories in a positive-psychology and motivational interviewing intervention for people with type 2 diabetes. Health Psychol Behav Med. 2022 Aug 4;10(1):713-730. doi: 10.1080/21642850.2022.2104724. eCollection 2022. PMID 35957957
- [Derived] Zambrano J, Celano CM, Chung WJ, Massey CN, Feig EH, Millstein RA, Healy BC, Wexler DJ, Park ER, Golden J, Huffman JC. Exploring the feasibility and impact of positive psychology-motivational interviewing interventions to promote positive affect and physical activity in type 2 diabetes: design and methods from the BEHOLD-8 and BEHOLD-16 clinical trials. Health Psychol Behav Med. 2020;8(1):398-422. doi: 10.1080/21642850.2020.1815538. Epub 2020 Sep 14. PMID 33763296
- [Derived] Feig EH, Harnedy LE, Celano CM, Huffman JC. Increase in Daily Steps During the Early Phase of a Physical Activity Intervention for Type 2 Diabetes as a Predictor of Intervention Outcome. Int J Behav Med. 2021 Dec;28(6):834-839. doi: 10.1007/s12529-021-09966-0. Epub 2021 Feb 11. PMID 33575971